CLINICAL TRIAL: NCT00967876
Title: Coronary Artery Stent Evaluation With 320-slice Computed Tomography - The CArS 320 Study
Acronym: CARS-320
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marc Dewey, PD, Charite University, Berlin, Germany
Other Study IDs: EA1/133/08
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Stenosis
Keywords: Men or women of any ethnic group scheduled to undergo conventional coronary angiography for suspected coronary artery stent stenosis
MeSH Terms: conditions — Coronary Stenosis; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The investigators aim at analyzing the diagnostic accuracy of 320-row CT for coronary stents.

ELIGIBILITY:
Inclusion Criteria:

* Suspected coronary artery in-stent restenoses based on clinical findings or findings on other noninvasive imaging tests and planned coronary angiography within the next 14 days.
* Able to understand and willing to sign the Informed CF.

Exclusion Criteria:

* Creatinine of above 2.0 mg/dl
* Age below 40 years
* Women of child bearing potential (no hysterectomy, no menopause, or menopause since less than 12 months) must demonstrate a negative pregnancy test performed within 24 hours before CT.
* Resting heart rate above 70 beats per minute and contraindications to beta blockers (e.g. moderate to severe bronchospastic disease, asthma)
* Atrial fibrillation, uncontrolled tachycardia, A-V block II or III degree or other non-sinus rhythms
* Inability to hold the breath for 10 seconds
* Hypotension < 80 mmHg systolic
* Unstable angina pectoris, acute myocardial infarction < 48h
* Continuous therapy with Dipyridamol
* Severe aortic stenosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent coronary artery stent placement in the past and are clinically indicated to undergo conventional coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, MD, PhD, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Zimmermann E, Dewey M. Whole-heart 320-row computed tomography: reduction of radiation dose via prior coronary calcium scanning. Rofo. 2011 Jan;183(1):54-9. doi: 10.1055/s-0029-1245629. Epub 2010 Aug 19. PMID 20725881
- [Background] Dewey M, Zimmermann E, Deissenrieder F, Laule M, Dubel HP, Schlattmann P, Knebel F, Rutsch W, Hamm B. Noninvasive coronary angiography by 320-row computed tomography with lower radiation exposure and maintained diagnostic accuracy: comparison of results with cardiac catheterization in a head-to-head pilot investigation. Circulation. 2009 Sep 8;120(10):867-75. doi: 10.1161/CIRCULATIONAHA.109.859280. Epub 2009 Aug 24. PMID 19704093
- [Background] Dewey M. Coronary CT versus MR angiography: pro CT--the role of CT angiography. Radiology. 2011 Feb;258(2):329-39. doi: 10.1148/radiol.10100161. No abstract available. PMID 21273517
- [Result] Rief M, Zimmermann E, Stenzel F, Martus P, Stangl K, Greupner J, Knebel F, Kranz A, Schlattmann P, Laule M, Dewey M. Computed tomography angiography and myocardial computed tomography perfusion in patients with coronary stents: prospective intraindividual comparison with conventional coronary angiography. J Am Coll Cardiol. 2013 Oct 15;62(16):1476-85. doi: 10.1016/j.jacc.2013.03.088. Epub 2013 Jun 19. PMID 23792193
- [Derived] Preuss D, Garcia G, Laule M, Dewey M, Rief M. Myocardial CT perfusion imaging for the detection of obstructive coronary artery disease: multisegment reconstruction does not improve diagnostic performance. Eur Radiol Exp. 2022 Jan 31;6(1):5. doi: 10.1186/s41747-021-00256-8. PMID 35099638
- [Derived] Rief M, Feger S, Martus P, Laule M, Dewey M, Schonenberger E. Acceptance of Combined Coronary CT Angiography and Myocardial CT Perfusion versus Conventional Coronary Angiography in Patients with Coronary Stents--Intraindividual Comparison. PLoS One. 2015 Sep 1;10(9):e0136737. doi: 10.1371/journal.pone.0136737. eCollection 2015. PMID 26327127
- [Derived] Feger S, Rief M, Zimmermann E, Martus P, Schuijf JD, Blobel J, Richter F, Dewey M. The Impact of Different Levels of Adaptive Iterative Dose Reduction 3D on Image Quality of 320-Row Coronary CT Angiography: A Clinical Trial. PLoS One. 2015 May 6;10(5):e0125943. doi: 10.1371/journal.pone.0125943. eCollection 2015. PMID 25945924